CLINICAL TRIAL: NCT00872118
Title: Brief Intervention for Socially Anxious Alcohol Abusers
Brief Title: Brief Intervention for Socially Anxious College Drinkers
Acronym: BISAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Giao Q. Tran, Ph.D., University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIAAA-Tran-AA014014; R21AA017291 (NIH); NIH Grant R21AA014014
Record Dates: First submitted 2009-03-27; First posted 2009-03-31 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Alcohol Consumption; Alcohol Negative Consequences; Social Anxiety
Keywords: alcohol consumption; social anxiety; brief intervention; motivational interviewing; cognitive behavioral
MeSH Terms: conditions — Alcohol Drinking | interventions — Crisis Intervention; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Brief Intervention for Socially Anxious Drinkers
  Interventions: Behavioral: Brief Intervention for Socially Anxious Drinkers (BISAD)
- 2 (Active Comparator): Enhanced Alcohol Skills and Education Program
  Interventions: Behavioral: Enhanced Alcohol Skills Building and Education Program

INTERVENTIONS:
Behavioral: Brief Intervention for Socially Anxious Drinkers (BISAD) — integrated alcohol and social anxiety individual intervention
  Arms: 1
Behavioral: Enhanced Alcohol Skills Building and Education Program — alcohol-focused group intervention
  Arms: 2

SUMMARY:
The purpose of this study is to develop and test a new brief intervention to reduce heavy drinking and social anxiety in college drinkers.

DETAILED DESCRIPTION:
Episodic alcohol abuse is common among college students. Recently, brief interventions focusing on motivational strategies and behavior skills to reduce heavy drinking and alcohol-related problems have shown beneficial small to medium effects in college drinkers who reported heavy drinking and/or alcohol-related problems. Most interventions have not taken into account psychiatric comorbidity, in particular social anxiety, a frequent problem for college students that has been linked to excessive alcohol use. This project will extend knowledge on brief interventions by integrating cognitive-behavioral therapeutic strategies for social anxiety with an existing alcohol intervention designed for college students.

The efficacy of a new integrated treatment, the Brief Intervention for Socially Anxious Drinkers (BISAD) was developed and tested. All participants reported heavy alcohol use, alcohol-related problems and social anxiety based on standardized measures. Phase I of the study focused on the development of the treatment manuals and measures of therapy integrity for BISAD and an alcohol-focused intervention, a modified treatment-as-usual at the local university. During this phase therapists were trained to administer the manualized interventions to study participants (N=12). Phase II included further refinement of the therapy integrity measures and data collection for the pilot study (N=41). Participants were randomized to either BISAD (n=21) or a modified treatment-as-usual (n=20) condition. The pilot study provide preliminary data on the efficacy of the proposed intervention in reducing heavy drinking, social anxiety, and their negative consequences at 1-month and 4-month follow-ups after treatment termination. These data provide estimated effect sizes for future testing of BISAD in a full-scale clinical trial. Furthermore, the study results contribute to the conceptualization and methodological development of combined interventions for other substance use and psychiatric problems.

ELIGIBILITY:
Inclusion Criteria:

1. at least one heavy drinking episode (4 or more drinks for women and 5 or more for men)
2. occasional to frequent drinking related problems
3. moderate social anxiety symptoms

Exclusion Criteria:

1. history of schizophrenia, bipolar disorder, organic brain syndrome or mental retardation
2. current illicit substance dependence, severe alcohol dependence, anxiety disorders (except simple phobia), unipolar depression, major medical illness, pregnancy, suicidality, or homicidality

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
heavy drinking days | pre-treatment, 1-month follow-up and 4-month follow-up
total alcohol consumption | pre-treatment, 1-month follow-up and 4-month follow-up
drinking-related negative consequences | pre-treatment, 1-month follow-up and 4-month follow-up
social (interactional) anxiety | pre-treatment, 1-month follow-up and 4-month follow-up

SECONDARY OUTCOMES:
alcohol expectancies of social evaluative situations | pre-treatment, 1-month follow-up and 4-month follow-up
drink refusal self-efficacy in social situations | pre-treatment, 1-month follow-up and 4-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Giao Q. Tran, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- Psychology Department, University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Tran, G.Q. (2008). Efficacy of a brief intervention for college hazardous drinkers with social anxiety: A randomized controlled pilot study. Alcoholism: Clinical and Experimental Research, 32 (Supplement), 190A.
- [Background] Tran, G.Q., Lanman, S.A., Perciful, M.S., Thompson, R.D., & Smith, J.P. (2006). Promising inexpensive methods for recruiting college-age heavy drinkers for brief alcohol and social anxiety interventions. Alcoholism: Clinical and Experimental Research, 30 (Supplement), 101A.